CLINICAL TRIAL: NCT07048431
Title: Evaluation of Chemotherapy-Induced Neuropathic Pain Using Shear Wave Elastography Measurements of the Tibial Nerve
Brief Title: Tibial Nerve Elastography in Chemotherapy-Induced Neuropathic Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Turan, MD, Principal Investigator, Ankara Etlik City Hospital
Other Study IDs: Tibial Nerve Elastography
Record Dates: First submitted 2025-06-21; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Tibial Neuropathy
Keywords: Chemotherapy-induced Peripheral Neuropathy; Tibial Neuropathy
MeSH Terms: conditions — Tibial Neuropathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chemotherapy-Induced Tibial Neuropathy Group: This group includes adult patients diagnosed with peripheral tibial neuropathy attributed to chemotherapy treatment. Participants must exhibit clinical signs or symptoms consistent with tibial nerve involvement, such as distal lower limb pain, paresthesia, weakness, or altered sensation in the tibial nerve distribution.
  Interventions: Diagnostic Test: Shear Wave Elastography Measurement
- Healthy Volunteers Group: This group consists of adult participants with no known acute or chronic medical conditions, neurological disorders, or history of chemotherapy or neurotoxic drug exposure. Individuals must be in good general health, as determined by medical history, physical examination. This group serves as a control population to establish baseline measurements.
  Interventions: Diagnostic Test: Shear Wave Elastography Measurement

INTERVENTIONS:
Diagnostic Test: Shear Wave Elastography Measurement — It is a non-invasive imaging technique used to evaluate tissue stiffness. This method involves the use of ultrasound-based shear wave elastography to assess bilateral tibial nerve, by measuring the speed of shear wave propagation through the tissue. Stiffness values are expressed in kilopascals (kPa).

SUMMARY:
This observational study aims to evaluate the tibial nerve stiffness using Shear Wave Elastography (SWE) in patients with chemotherapy-induced peripheral neuropathy (CIPN) compared to healthy volunteers. A total of 25 patients with a DN4 score ≥4 and 25 healthy controls will be assessed. Parameters including nerve diameter, cross-sectional area, depth, and shear wave velocity (V value) will be measured. Demographic and clinical data such as age, gender, chemotherapy protocol, duration, comorbidities, and medications will also be collected. The goal is to investigate SWE as a non-invasive diagnostic tool for CIPN by identifying differences in nerve elasticity between groups.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common dose-limiting side effect observed in 30-40% of patients receiving neurotoxic chemotherapy. CIPN typically presents with sensory symptoms such as paresthesia, numbness, balance disturbances, heightened pain sensitivity, and deep tendon reflex loss. The severity and progression of neuropathy vary widely among patients.

The diagnosis of peripheral neuropathy is based on clinical symptoms and is often supported by nerve conduction studies such as electromyography (EMG). However, EMG can be time-consuming and may be insufficient in advanced cases due to loss of nerve action potentials. Furthermore, subclinical cases of neuropathy may go undetected by EMG.

Recent evidence suggests that pathophysiological changes in CIPN may lead to increased nerve stiffness. Shear Wave Elastography (SWE), a non-invasive ultrasound-based technique, allows for quantitative evaluation of tissue elasticity by measuring shear wave velocity (V value in m/s) and calculating stiffness (E value in kPa). Unlike strain elastography, SWE does not require manual compression, making it more objective and reproducible.

This observational, case-control study aims to assess tibial nerve elasticity using SWE in patients diagnosed with CIPN and to compare the findings with healthy controls. A total of 25 patients with CIPN (defined as a DN4 score ≥4) and 25 age-matched healthy volunteers without neuropathy symptoms will be included. All participants will undergo ultrasound and SWE measurements of bilateral tibial nerve.

Parameters recorded will include the anteroposterior and lateral-medial diameter, cross-sectional area, distance from the skin, and the mean shear wave velocity (V value) obtained from three repeated measurements. In addition, demographic and clinical data such as age, gender, chemotherapy protocol and duration, comorbidities, and current medications will be collected.

The primary objective is to investigate whether tibial nerve elasticity differs significantly between CIPN patients and healthy individuals. This study aims to explore SWE as a potential supportive diagnostic tool for early detection or monitoring of CIPN.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* DN4 score ≥4
* Anatomical suitability for tibial nerve ultrasound and SWE assessment
* Providing written informed consent

Exclusion Criteria:

* Presence of diabetes mellitus
* Alcohol use
* Polyneuropathy due to genetic or toxic causes
* Fracture, skin lesion, or edema in the lower extremity
* Severe systemic diseases (e.g., liver, kidney, heart, or lung)
* Inability to visualize the tibial nerve anatomically
* Cognitive or psychiatric disorders preventing cooperation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study included adults aged 18-75 years, divided into two groups: 25 patients with chemotherapy-induced peripheral neuropathy (CIPN) and DN4 scores ≥4, and 25 healthy controls without neuropathy symptoms. All participants underwent clinical screening and were anatomically suitable for tibial nerve ultrasound and shear wave elastography (SWE). Both tibial nerves were evaluated in each subject. Individuals with diabetes mellitus, alcohol use, genetic or toxic neuropathies, systemic diseases, lower limb trauma or lesions, or cognitive/psychiatric disorders affecting cooperation were excluded. The goal was to ensure a homogeneous population for accurate elastographic comparison.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Shear Wave Elastography (SWE) Stiffness Value | Single SWE measurement performed within the first week of study inclusion
  Shear Wave Elastography (SWE) is an imaging technique used to quantify tissue stiffness by measuring the propagation speed (V, m/s) of shear waves and converting it into elasticity values (E, kilopascals, kPa). Higher values may indicate fibrosis or increased tension, while lower values may reflect fatty infiltration or atrophy. In peripheral nerves, SWE has been used to assess elasticity in neuropathic conditions. Research shows that affected nerves in neuropathy exhibit increased stiffness compared to healthy nerves. Both shear wave velocity (V) and elasticity modulus (E) can be measured, offering objective, quantitative data to detect and monitor structural nerve changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Etlik, Turkey (Türkiye)